CLINICAL TRIAL: NCT07184619
Title: A Phase III, 12-week, Prospective, Randomized, Double-blind, Placebo-controlled, Parallel-group, Multi-center Study to Determine the Efficacy, Safety, and Tolerability of a Dose of 15 mg Bid of Evenamide as add-on in Patients With Documented Treatment-resistant Schizophrenia, Which is Not Adequately Controlled by a Stable Therapeutic Dose of the Patient's Current Antipsychotic Medication(s)
Brief Title: Evenamide, a Glutamate Release Modulator, as Add-On to Standard of Care in Subjects With Documented Treatment-Resistant Schizophrenia
Acronym: ENIGMA-TRS 2
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Newron Pharmaceuticals SPA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NW-3509/022/III/2024
Record Dates: First submitted 2025-09-18; First posted 2025-09-22 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Treatment-resistant Schizophrenia
Keywords: evenamide; treatment-resistant schizophrenia; antipsychotic; schizophrenia; TRS; add-on treatment
MeSH Terms: conditions — Schizophrenia, Treatment-Resistant; Schizophrenia | interventions — BID protein, human

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Evenamide 15 mg bid (Experimental): Evenamide capsules 15 mg bid for a total of 12 weeks of add-on treatment
  Interventions: Drug: Evenamide 15 mg bid
- Placebo (Placebo Comparator): Matching placebo capsules bid for a total of 12 weeks of add-on treatment
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Evenamide 15 mg bid — Evenamide capsules 15 mg bid for a total of 12 weeks of add-on treatment
  Arms: Evenamide 15 mg bid
Drug: Placebo — Matching placebo capsules bid for a total of 12 weeks of add-on treatment
  Arms: Placebo

SUMMARY:
This is a prospective, 12-week, randomized, double-blind, placebo-controlled study, designed to evaluate the efficacy, safety, and tolerability of a dose of evenamide of 15 mg bid, compared to placebo, as add-on treatment in patients with documented treatment-resistant schizophrenia (TRS) who have prospectively demonstrated inadequate response to their current stable therapeutic dose of an antipsychotic(s). Approximately 400 patients will be randomized equally (1:1) to each of the two treatment groups in this study.

ELIGIBILITY:
Key Inclusion Criteria:

* Age - 18 years, or older.
* If female, the subject has a negative pregnancy test at the screening visit and at baseline, is not lactating, and agrees to use adequate contraception, unless not of childbearing potential.
* Meets current DSM-5-TR criteria for schizophrenia.
* Has shown treatment-resistance to antipsychotics as per TRRIP working group definition (Howes et al., 2017).
* Currently receiving "standard of care" therapy of a minimal recommended therapeutic dose of one or more antipsychotic(s).
* Has a Clinical Global Impression - Severity of disease (CGI-S) rating of "mildly ill" to "among the most extremly ill" at baseline.
* Has a BPRS total score ≥ 45 at screening and baseline.
* Has a PANSS total score ≥ 70 at baseline.
* Has a Global Assessment of Functioning (GAF) scale total score ≤ 50.
* Adherence to prescribed antipsychotic treatment.
* Patient has provided written informed consent prior to participating in the study.

Key Exclusion Criteria:

* Current DSM-5-TR diagnosis of schizophreniform disorder, schizoaffective disorder, or other primary psychiatric diagnosis, such as bipolar disorder or major depressive disorder
* History (within three months of study entry) or current diagnosis of "Substance Use Disorder" as defined by the DSM-5-TR criteria.
* Severity of current episode of psychosis requires that the patient be hospitalized to stabilize the severity of his/her psychotic symptoms. However, these patients may qualify for the study provided their antipsychotic dose has been stable for 6 weeks prior to screening.
* History or current diagnosis of other psychiatric or behavioral disorders.
* Known suicidal risk, or a suicide attempt within the past 2 years.
* History of neuroleptic malignant syndrome or priapism.
* Disease/medical condition of any type that may impact the patient's safety or interfere with any of the study evaluations.
* History or current diagnosis of epilepsy or seizure disorder, or occurrence of a seizure within the past year, or repeated drug-induced seizures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2026-01-23 (Actual); Primary Completion 2026-09-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Change from baseline to endpoint (Week 12) on the total score of the Positive and Negative Syndrome Scale (PANSS). | From Baseline to Week 12
  Efficacy measured by the mean change from baseline to endpoint of Positive and Negative Syndrome Scale [PANSS] total score: a 30-item scale that was designed to assess various symptoms of schizophrenia each rated on a 7-point scale that ranges from 1 (absent) to 7 (extreme psychopathology).
Incidence of treatment-emergent adverse events (TEAEs), AEs leading to discontinuation (ADOs), and serious AEs (SAEs). | From Baseline to 30-day Safety Follow up (12 Weeks of treament + 30-day safety follow up)
  Safety and tolerability of a dose of evenamide of 15 mg bid, compared to placebo. The assessment of safety and tolerability will be based primarily on the incidence of treatment-emergent adverse events (TEAEs), AEs leading to discontinuation (ADOs), and serious AEs (SAEs).

SECONDARY OUTCOMES:
Change from baseline to endpoint (Week 12) on the Clinical Global Impression - Severity of illness (CGI-S) score. | From Baseline to Week 12
  Efficacy measured by the mean change from baseline to endpoint on the Clinical Global Impression Severity of Illness (CGI-S) scale: a 7-point scale ranging from 1 (no symptoms) to 7 (very severe) to assess the severity of a subject's condition.
Proportion of patients rated as 'improved' on the CGI-C at endpoint (Week 12). | Week 12
  Efficacy measured by Clinical Global Impression of Change [CGI-C]: a 7-point scale, ranging from 1 (very much improved) to 7 (very much worse), with a score of 4 indicating "no change". Patients with ratings of 1,2 or 3 are considered as 'improved'.
Change from baseline to endpoint (Week 12) on the Positive Symptoms sub-scale score of the PANSS. | From Baseline to Week 12
  Efficacy measured by the mean change from baseline to endpoint on the Positive subscale score of the PANSS: a 7-item subscale designed to assess positive symptoms of schizophrenia each rated on a 7-point scale that ranges from 1 (absent) to 7 (extreme psychopathology).
Change from baseline to endpoint (Week 12) on the Personal and Social Performance (PSP) scale. | From Baseline to Week 12
  Efficacy measured by the mean change from baseline to endpoint on the PSP scale: a 100-point single-item rating scale subdivided into 10 equal intervals that designed to assess the routine social functioning of patients with psychiatric disorders.
Change from baseline to endpoint (Week 12) on the Quality of Life Enjoyment and Satisfaction Questionnaire - Short Form scale (Q-LES-Q-SF). | From Baseline to Week 12
  Efficacy measured by the mean change from baseline to endpoint on the total score of the Quality of Life Enjoyment and Satisfaction Questionnaire: a 16-item scale, each rated from 1 (very poor) to 5 (very good).

OTHER OUTCOMES:
Change from baseline to endpoint (Week 12) on the Negative Symptoms sub-scale score of the PANSS. | From Baseline to Week 12.
  Efficacy measured by the mean change from baseline to endpoint on the Positive subscale score of the PANSS: this is a 7-item subscale that was designed to assess negative symptoms of schizophrenia each rated on a 7-point scale that ranges from 1 (absent) to 7 (extreme psychopathology).
Change from baseline to endpoint (Week 12) on the Calgary Depression Scale for Schizophrenia (CDSS). | From Baseline to Week 12
  Efficacy measured by the mean change from baseline to endpoint on the CDSS: a 9-item, observer-rated, semi-structured, goal-directed interview, validated for diagnosing depression in patients with schizophrenia. Each item is scored between "Absent" (0) to "Severe" (3), based on operational criteria.
Change from baseline to endpoint (Week 12) on the Global Assessment of Functioning (GAF) scale. | From Baseline to Week 12.
  Efficacy measured by the mean change from baseline to endpoint on the GAF scale ranging from 0 (inadequate information) to 100 (superior functioning), and is divided into 10-point ranges of functioning.
Change from baseline to endpoint (Week 12) on the Medication Satisfaction Questionnaire (MSQ). | From Baseline to Week 12
  Efficacy measured by the mean change from baseline to endpoint on the Medication Satisfaction Questionnaire (MSQ) which is a single-item, 7-point scale for patients with schizophrenia to rate their satisfaction with their antipsychotic medication ranging from "extremely dissatisfied" (1) to "extremely satisfied" (7).
Change from baseline to endpoint (Week 12) on the Cognitive Test Battery. | From Baseline to Week 12
  Efficacy measured by the mean change from baseline on the scores of the Cognitive Test Battery. This includes: the Digit Symbol Substitution test, Trail Making Test (Parts A and B), d2 Test of Attention, and verbal fluency measures.

CONTACTS AND LOCATIONS:
Overall Officials: Ravi Anand, MD, Study Director — Newron Pharmaceuticals
Locations (5):
- United States (5):
  - UCLA DGSOM, UCLA Health, UCLA Semel Institute, Los Angeles, California
  - University of Miami, Miller School of Medicine; Jackson Behavioral Health Hospital, Miami, Florida
  - Grady Behavioral Health Center, -Department of Psychiatry and Behavioral Sciences, Emory University School of Medicine, Atlanta, Georgia
  - Department of Psychiatry and Behavioral Sciences, Johns Hopkins University School of Medicine, Baltimore, Maryland
  - Manhattan Psychiatric Center, The Nathan Kline Institute for Psychiatric Research, New York, New York

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Anand R, Turolla A, Chinellato G, Sansi F, Roy A, Hartman R. Efficacy and safety of evenamide, a glutamate modulator, added to a second-generation antipsychotic in inadequately/poorly responding patients with chronic schizophrenia: Results from a randomized, double-blind, placebo-controlled, phase 3, international clinical trial. Neuropharmacology. 2025 Mar 15;266:110275. doi: 10.1016/j.neuropharm.2024.110275. Epub 2024 Dec 19. PMID 39708914
- [Background] Anand R, Turolla A, Chinellato G, Roy A, Hartman RD. Therapeutic Effect of Evenamide, a Glutamate Inhibitor, in Patients With Treatment-Resistant Schizophrenia (TRS): Final, 1-Year Results From a Phase 2, Open-Label, Rater-Blinded, Randomized, International Clinical Trial. Int J Neuropsychopharmacol. 2024 Dec 28;28(1):pyae061. doi: 10.1093/ijnp/pyae061. PMID 39661380
- [Background] Anand R, Turolla A, Chinellato G, Roy A, Hartman RD. Phase 2 Results Indicate Evenamide, A Selective Modulator of Glutamate Release, Is Associated With Clinically Important Long-Term Efficacy When Added to an Antipsychotic in Patients With Treatment-Resistant Schizophrenia. Int J Neuropsychopharmacol. 2023 Aug 29;26(8):523-528. doi: 10.1093/ijnp/pyad035. PMID 37349110